CLINICAL TRIAL: NCT04121507
Title: A Prospective Phase II Clinical Study to Assess the Efficacy and Toxicity of High-dose Chemotherapy Followed by Allogeneic Stem Cell Transplantation as Treatment of Primary Progressive and Relapsed Aggressive Non-Hodgkin Lymphoma
Brief Title: ASTRAL- a Clinical Study to Assess the Efficacy and Toxicity of High-dose Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GWT-TUD GmbH (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ASTRAL / GLA-aNHL-R1
Record Dates: First submitted 2019-07-31; First posted 2019-10-10 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2022-04

CONDITIONS: Aggressive Non-hodgkin Lymphoma (aNHL); Lymphoma, B-Cell; Lymphoma, T-Cell
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, T-Cell | interventions — fludarabine; Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- alloSCT (Experimental): defined high-dose chemotherapy (HDT) followed by allogeneic stem cell transplantation (alloSCT)
  Interventions: Drug: High dose chemotherapy before allogeneic stem cell transplantation (alloSCT); Procedure: Bone marrow histology; Diagnostic Test: clinical and laboratory parameters; Diagnostic Test: PET-CT or CT

INTERVENTIONS:
Drug: High dose chemotherapy before allogeneic stem cell transplantation (alloSCT) — High-dose therapy (HDT) prior to alloSCT will consist of FTC
  Other Names: fludarabine, thiotepa ,cyclophosphamide (FTC)
Procedure: Bone marrow histology — Bone marrow histology at staging and restaging is only mandatory if the bone marrow was initially involved
Diagnostic Test: clinical and laboratory parameters — During staging and restaging examinations, all clinical and laboratory parameters relevant for therapy.
Diagnostic Test: PET-CT or CT — Metabolic CR in a PET-CT scan after the last cycle of therapy prior to planned SCT. Consists preferably of a PET-CT or a CT scan according to local practice and other appropriate diagnostic procedures with respect to the sites of primary involvement.

SUMMARY:
A prospective Phase II clinical study to assess the efficacy and toxicity of high dose chemotherapy (HDT) followed by allogeneic stem cell transplantation (allo- or autoSCT) as treatment of primary progressive and relapsed aggressive Non-Hodgkin Lymphoma (NHL) - ASTRAL

DETAILED DESCRIPTION:
This is a clinical study to assess the treatment (efficacy and toxicity) with a high dosed chemotherapy followed by stem cell transplantation in patients suffering from primary progressive and relapsed aggressive Non-Hodgkin Lymphoma (NHL)

After end of the active study phase, patients will receive further standard medical care at the discretion of the treating physician. The clinical consultants will provide advice on further treatment if requested.

ELIGIBILITY:
Inclusion Criteria:

Subjects must fulfill all of the following criteria to be included in this trial:

1. Provision of written informed consent and specifically the consent to the collection and processing of health-related data
2. Age: 18 years and older
3. Gender: Male and female patients
4. Histology
5. Diagnosis of relapsed or primary progressive aggressive B- or T-cell lymphoma including:

   1. B-Cell non-hodgkin lymphoma (B-NHL) or
   2. T-Cell non-hodgkin lymphoma (T-NHL):
6. Staging at relapse or progression (data should not be older than 4 weeks):
7. Staging after 2 or 3 cycles of salvage treatment:
8. Donor availability:
9. Females of childbearing potential (FCBP) must:

   * Understand the potential teratogenic risk to the unborn child
   * Understand the need and agree to utilize two reliable forms of contraception
   * Understand and agree to inform the investigator if a change or stop of method of contraception is needed
   * Be capable of complying with effective contraceptive measures
   * Be informed and understand the potential consequences of pregnancy and the need to notify her study doctor immediately if there is a risk of pregnancy
   * Understand the need to commence the study treatment as soon as study drug is dispensed following a negative pregnancy test
   * Understand the need and accept to undergo pregnancy testing based on the frequency outlined in this protocol
   * Agree to abstain from breastfeeding during study participation
10. Males must:

    * Agree to use a latex condom during any sexual contact with females of childbearing potential
    * Agree to refrain from donating semen or sperm while on the study drugs and should seek for sperm cryopreservation before therapy is started and should not father a child while treated and during one year after end of study treatment
11. Females of non-childbearing potential:

Exclusion Criteria:

Subjects are to be excluded from the study if they display any of the following criteria:

1. Pregnant females; lactating women must end breast feeding before start of study treatment
2. Serious accompanying disorder or impaired organ function
3. Central nervous system (CNS) involvement of lymphoma - to be examined in case of clinical symptoms
4. History of severe cardiac diseases, and cardiac function impairment
5. Severe kidney disease
6. HIV-positivity
7. Hepatitis B and C as defined by seropositivity
8. Patients under legal guardianship regarding medical decisions
9. Ongoing treatment or study procedures within any other clinical trial with the exception of follow up
10. Ongoing exclusion periods of other clinical studies after end of treatment
11. In patients tested: Metabolic Computer tomography (CR) in a positron emission tomography-Computer tomography (PET-CT) scan after the last cycle of therapy prior to planned SCT
12. Subjects with known hypersensitivity to the study drugs
13. Criteria which in the opinion of the investigator precluded participation for scientific reasons, for reasons of compliance, or for reasons of the subject's safety
14. Commitment to an institution by virtue of an order issued either by the judicial or the administrative authorities
15. Dependency on the sponsor, trial site or investigator
16. Additional exclusion criteria with respect to summary of product characteristics (SmPC) of the investigational medical product (IMPs) fludarabine, thiotepa, cyclophosphamide:

    1. Known hypersensitivity to fludarabine, thiotepa, cyclophosphamide or one of their metabolites
    2. Renal impairment
    3. Decompensated haemolytic anaemia
    4. Concurrent application of vital vaccines
    5. Cystitis
    6. Renal tract obstruction
    7. Active and uncontrolled infection
    8. Notice: myelosuppression and impaired hematopoietic function is not an exclusion criterion as this usual contraindication to the application to any of the IMPs will be overcome by the stem cell transplantation following conditioning therapy.

       -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2023-02-02 (Actual)

PRIMARY OUTCOMES:
Measurement of efficacy variables, Rate of Progression free survival (PFS) | 1 year after SCT
  To compare a defined high dose therapy (HDT) with study medication followed by alloSCT lead to treatment results in terms of PFS, that are better than results obtained with high-dose therapy and autoSCT in a comparable Patient Population ( historical data).

SECONDARY OUTCOMES:
Measurement of efficacy variables, Rate of complete remissions (CR) | 1 year after stem cell transplantation (SCT)
  Number of complete remissions divided by the number of patients (CR),
Measurement of efficacy variables, Rate of partial remissions (PR) | 1 year after SCT
  Number of partial remissions divided by the number of patients (PR);
Measurement of efficacy variables, Rate of complete and partial remissions (ORR) | 1 year after SCT
  Number of complete and partial remissions divided by the number of patients (ORR);
Measurement of efficacy variables, Rate of progressive diseases (PD) | 1 year after SCT
  Number of progressive diseases after SCT divided by the number of patients (PD);
Measurement of efficacy variables, Rate of relapse (RR) | 1 year after SCT
  safety item
Measurement of efficacy variables, Rate of treatment-related mortality | 1 year after SCT
  treatment-related death divided by the number of patients
Rate of event free survival at 1 year (EFS) | 1 year after SCT
  safety item
Measurement of efficacy variables, Rate of overall survival at 1 year (OS) | 1 year after SCT
  safety item
Measurement of efficacy variables, Rate of non-relapse mortality (NRM) | 1year after SCT
  safety item
Measurement of efficacy variables, Causes of death | 1year after SCT
  safety item
Measurement of efficacy variables, Incidence and severity of acute and chronic graft versus host disease (GvHD); | until the last Follow-Up Visit ( 1-2 Year after SCT)
  safety item
Measurement of efficacy variables, Adverse events (AEs) grade 3 and 4 | until about day 100 after SCT.
  safety item
Measurement of efficacy variables, Serious adverse events (SAEs) | until about day 100 after SCT.
  safety item
Measurement of number of blood cells | 1year after SCT
  recovery of White blood cells and platelets
Measurement of efficacy variables, Rate of infections | 1year after SCT
  safety item

CONTACTS AND LOCATIONS:
Overall Officials: Bertram Glass, Prof. Dr., Principal Investigator — Helios Klinikum Berlin-Buch
Locations (13):
- Germany (13):
  - HELIOS Klinik Berlin-Buch, Klinik für Hämatologie und Stammzelltransplantation, Berlin, Brandenburg
  - Klinikum Augsburg, Medizinische Klinik II, Augsburg
  - Medizinisches Universitätsklinikum, Bochum
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Universitätsklinikum Carl Gustav Carus Dresden, Medzinische Klinik I, Dresden
  - Universitäsklinikum Düsseldorf, Düsseldorf
  - Universitätsmedizin Göttingen Klinik für Hämatologie/Med. Onkologie, Göttingen
  - Universitätsklinikum Halle, Halle
  - Universitätsklinikum Hamburg-Eppendorf, Zentrum für Onkologie, Interdisziplinäre Klinik und Poliklinik für Stammzelltransplantation, Hamburg
  - Universitätsklinikum Heidelberg, Medizinische Klinik, Innere Medizin V, Heidelberg
  - Universitätsklinikum Jena, Klinik für Innere Medizin, Abtl. Hämatologie und Innternistische Onkologie, Jena
  - Universitätsklinikum Münster, KMT-Zentrum/ Med. Klinik A, Münster
  - Klinikum Stuttgart, Stuttgart

IPD SHARING:
Plan to Share IPD: No